CLINICAL TRIAL: NCT00443820
Title: A Randomized, Double-blind, Vehicle-controlled, Multicenter, Parallel Group Study to Assess the Efficacy, Safety, and Tolerability of Topical Terbinafine Hydrogen Chloride (HCl) Formulation for 24 or 48 Weeks of Treatment in Patients With Mild to Moderate Toenail Onychomycosis
Brief Title: Efficacy Safety, and Tolerability of Topical Terbinafine in Patients With Mild to Moderate Toenail Fungus of the Big Toenail
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSFO327N2302
Record Dates: First submitted 2007-03-02; First posted 2007-03-06 (Estimated); Results first posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-03

CONDITIONS: Onychomycosis
Keywords: Toenail fungus; Onychomycosis; Nail fungus; Toenail fungal infection; Tinea unguium; Dermatophytes; Foot dermatoses
MeSH Terms: conditions — Onychomycosis; Foot Dermatoses | interventions — Terbinafine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis (NSO) for 48 weeks
  Interventions: Drug: terbinafine
- 2 (Placebo Comparator): Vehicle (placebo) for 48 weeks
  Interventions: Drug: Placebo
- 3 (Experimental): Terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis (NSO) for 24 weeks
  Interventions: Drug: terbinafine
- 4 (Placebo Comparator): Vehicle (placebo) for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: terbinafine — Terbinafine hydrochloride (HCl) 10 % nail solution for onychomycosis (NSO) once daily for 48 weeks
  Other Names: Lamisil
  Arms: 1
Drug: Placebo — Vehicle (placebo) once daily for 48 weeks
  Arms: 2
Drug: terbinafine — Terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis once daily for 24 weeks
  Other Names: Lamisil
  Arms: 3
Drug: Placebo — Vehicle (placebo) once daily for 24 weeks
  Arms: 4

SUMMARY:
This study is designed to assess the efficacy, safety and tolerability of a topical formulation of terbinafine solution applied daily in patients with toenail fungus. This trial will study patients with mild to moderate toenail fungus disease of the big toenail and their responses to two treatment durations, 24 or 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and females 12 - 75 years of age
* Fungal toenail infection of one or both of the large (great) toenails
* The nail infection must be due to a dermatophyte, (mixed infections dermatophyte and non-dermatophyte] are not allowed)

Exclusion Criteria:

* Target foot must not have severe plantar (moccasin) tinea pedis that would require systemic therapy. Mild to moderate tinea pedis (athlete's foot) infection should be treated with terbinafine prior to baseline or at any time during the trial. Other topical treatments for athlete's foot may be recommended at the discretion of the investigator.
* Subjects must not have abnormalities of the nail that could prevent a normal appearing nail if clearing of infection is achieved
* No administration of systemic antifungal medications within 6 months prior to screening visit
* No application of prescription topical antifungal medications for toenail fungus within 3 months or other commercially available topical medications for toenail fungus applied directly to the toenails within 1 month prior to screening visit
* No professional pedicures or application of any nail polish product or nail cosmetic to the toenails after the screening visit
* Known pregnancy or lactation at time of enrollment

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2006-12; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (20):
  - Dr. Fred D. Youngswick, Novato, California
  - Dr. Larry Doehring, Northglenn, Colorado
  - Dr. Robert P. Dunne, Melbourne, Florida
  - Dr. Mark Ling, Newnan, Georgia
  - Dr. Jesse Plasencia, Chicago, Illinois
  - Dr. John Mallory, Overland Park, Kansas
  - Dr. Jeffrey Conrow, Topeka, Kansas
  - Dr.Michael Kaye, Covington, Louisiana
  - Dr. Max Weisfeld, Baltimore, Maryland
  - Dr. Linda Stein-Gold, Detroit, Michigan
  - Dr. Anna Glaser, St Louis, Missouri
  - Dr. Richard Scher, New York, New York
  - Dr. Joseph Jorrizo, Winston-Salem, North Carolina
  - Dr. Anne Lucky, Cincinnati, Ohio
  - Dr. Rich Phoebe, Portland, Oregon
  - Dr. Patricia Westmorland, Simpsonville, South Carolina
  - Dr. David Horowitz, Nashville, Tennessee
  - Dr. Jay Lifshen, Irving, Texas
  - Dr. Richard Pollak, San Antonio, Texas
  - Dr. Patrick Agnew, Virginia Beach, Virginia
- Novartis Investigative Site, Various Cities, France
- Germany (2):
  - Novartis, Investigative Site
  - Novartis Investigative Site, Various Cities

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This randomized, double -blind, vehicle -controlled, multicenter, parallel group study was designed to assess the efficacy, safety and tolerability of a topical formulation of terbinafine hydrogen chloride 10% topical solution (TTS10%) applied daily in patients with toenail onychomycosis. Started 07 DEC 2006 and ending 27 JUN 2008.
Groups:
- Terbinafine 24 Weeks: Terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis (NSO) for 24 weeks
- Vehicle 24 Weeks: Vehicle (placebo) for 24 weeks
- Terbinafine 48 Weeks: Terbinafine hydrochloride (HCl) 10 % Nail Solution for Onychomycosis (NSO) for 48 weeks
- Vehicle 48 Weeks: Vehicle (placebo) for 48 weeks
Period: Overall Study
Arm/Group | Terbinafine 24 Weeks | Vehicle 24 Weeks | Terbinafine 48 Weeks | Vehicle 48 Weeks
Started | 133 | 130 | 135 | 128
Safety Population | 131 (Participants who received study drug and had at least one post-baseline safety assessment.) | 129 | 134 | 126
Completed | 112 | 111 (A participant from this gr. discont'ed due to renal failure, was counted as an AE and also as a SAE.) | 117 | 111
Not Completed | 21 | 19 | 18 | 17
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Lack of Efficacy | 3 | 2 | 1 | 1
Not completed — Protocol Violation | 2 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 6 | 7 | 8 | 9
Not completed — Lost to Follow-up | 9 | 8 | 6 | 5
Not completed — Administrative problems | 0 | 0 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Terbinafine 24 Weeks | Vehicle 24 Weeks | Terbinafine 48 Weeks | Vehicle 48 Weeks | Total
Number analyzed (Participants) | 133 | 130 | 135 | 128 | 526
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 1 | 1
  Between 18 and 65 years | 93 | 103 | 95 | 97 | 388
  >=65 years | 40 | 27 | 40 | 30 | 137
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 39 | 41 | 35 | 149
  Male | 99 | 91 | 94 | 93 | 377

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Assessed by the Percentage of Participants With Complete Cure at the End of Study (Week 52) After Treating for 24 or 48 Weeks
Description: Complete cure is defined as negative KOH microscopy and negative culture for dermatophytes and no residual involvement of the target toenail.
Time Frame: 52 weeks
Population: Intent to treat (ITT) population, Last observation carried forward (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Terbinafine 24 Weeks | Vehicle 24 Weeks | Terbinafine 48 Weeks | Vehicle 48 Weeks
Number analyzed (Participants) | 133 | 130 | 135 | 128
Percentage of participants | 1.50 [-1.82 to 3.29] | 0.77 [-1.82 to 3.29] | 2.96 [0.10 to 5.82] | 0 [0.10 to 5.82]

2. Secondary Outcome: Efficacy Assessed by the Percentage of Participants With Mycological Cure at the End of Study After Treating Participants for 24 or 48 Weeks
Description: Mycological cure is defined as negative KOH microscopy and negative culture for dermatophytes.
Time Frame: 52 weeks
Population: Intent to treat (ITT) population, Last observation carried forward (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Terbinafine 24 Weeks | Vehicle 24 Weeks | Terbinafine 48 Weeks | Vehicle 48 Weeks
Number analyzed (Participants) | 133 | 130 | 135 | 128
Percentage of participants | 15.04 [1.54 to 16.23] | 6.15 [1.54 to 16.23] | 22.22 [6.00 to 22.82] | 7.81 [6.00 to 22.82]

3. Secondary Outcome: Efficacy Assessed by the Percentage of Participants With Clinical Effectiveness at the End of Study After Treating Participants for 24 or 48 Weeks
Description: Clinical effectiveness is defined as negative KOH microscopy and negative culture for dermatophytes and <= 10% residual involvement of the target toenail.
  Clinical effectiveness was a composite binary variable defined as "Yes" if:
  * If mycological cure (negative KOH and negative culture for dermatophytes) and
  * = 10% residual involvement of the target toenail "No" if otherwise
Time Frame: 52 weeks
Population: Intent to treat (ITT) population, Last observation carried forward (LOCF)
Measure: Number; unit: Percentage of participants
Arm/Group | Terbinafine 24 Weeks | Vehicle 24 Weeks | Terbinafine 48 Weeks | Vehicle 48 Weeks
Number analyzed (Participants) | 133 | 130 | 135 | 128
Percentage of participants | 3.01 | 0.77 | 5.93 | 0.78

4. Secondary Outcome: Safety and Tolerability Assessed by the Number of Participants With Adverse Events
Description: Safety and tolerability data as assessed by the number of participants with Adverse Events (AE), Serious Adverse Events, Drug discontinuation due to an AE and death. Additional details can be found in the Adverse Event Section.
Time Frame: 52 weeks
Population: Safety Population
Measure: Number; unit: Number of participants
Arm/Group | Terbinafine 24 Weeks | Vehicle 24 Weeks | Terbinafine 48 Weeks | Vehicle 48 Weeks
Number analyzed (Participants) | 131 | 129 | 134 | 126
Number of participants
  At least 1 AE | 80 | 72 | 94 | 87
  At least 1 SAE | 8 | 3 | 9 | 7
  Study drug discontinued due to an AE | 0 | 1 | 1 | 0
  Death | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: 52 weeks
Description: Safety population consisting of all participants who had at least one dose of study drug and had at least one post-baseline safety assessment.
Arm/Group | Terbinafine 24 Weeks | Vehicle 24 Weeks | Terbinafine 48 Weeks | Vehicle 48 Weeks
Serious Adverse Events (participants affected / at risk) | 8/131 | 3/129 | 9/134 | 7/126
Other Adverse Events (participants affected / at risk) | 37/131 | 38/129 | 54/134 | 52/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Terbinafine 24 Weeks (N=131) | Vehicle 24 Weeks (N=129) | Terbinafine 48 Weeks (N=134) | Vehicle 48 Weeks (N=126)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Near drowning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 1
Bladder prolapse (Renal and urinary disorders) | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Micturition disorder (Renal and urinary disorders) | 0 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Terbinafine 24 Weeks (N=131) | Vehicle 24 Weeks (N=129) | Terbinafine 48 Weeks (N=134) | Vehicle 48 Weeks (N=126)
Influenza (Infections and infestations) | 2 | 1 | 13 | 10
Nasopharyngitis (Infections and infestations) | 13 | 11 | 15 | 15
Sinusitis (Infections and infestations) | 3 | 0 | 4 | 7
Upper respiratory tract infection (Infections and infestations) | 4 | 4 | 4 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7 | 6 | 12
Headache (Nervous system disorders) | 21 | 21 | 28 | 23
Hypertension (Vascular disorders) | 1 | 3 | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.